CLINICAL TRIAL: NCT03409354
Title: Tele-Rehabilitation Pilot Evaluation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Miho Asano, Assistant Professor, National University of Singapore
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MHHISDRFP16217
Record Dates: First submitted 2018-01-11; First posted 2018-01-24 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Fractures, Bone; Stroke; Lower Limb Joint Replacement (Hip or Knee); Lower Limb Amputation; Pneumonia; Fall; Deconditioning; Musculoskeletal Conditions (e.g., Tendinitis, Capsulitis)
MeSH Terms: conditions — Fractures, Bone; Stroke; Pneumonia; Tendinopathy; Bursitis | interventions — Telerehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-rehabilitation (Experimental): Tele-rehabilitation via iPad.
  Interventions: Behavioral: Tele-rehabilitation
- Usual care (Active Comparator): Usual rehabilitation care, prescribed by rehabilitation therapists at participating centers and performed by participants at participating centers.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Tele-rehabilitation — There are five different categories of exercise in the rehabilitation program, which combines both physiotherapy (Category 1 to 4) and occupational therapy components (Category 5). Each tele-therapy session could cover all five categories of exercises. Progression of levels within each exercise within each category should be determined by the tele-therapist and in consultation with the participant.
  Arms: Tele-rehabilitation
Behavioral: Usual care — Usual rehabilitation care (e.g., PT, OT and ST), prescribed by rehabilitation therapists at participating centers and performed by participants at participating centers.
  Arms: Usual care

SUMMARY:
A proof of concept randomized controlled trial (RCT) only evaluated the National University of Singapore's (NUS) T-Rehab tele-rehabilitation (TR) system at a home setting where rehabilitation was provided on an individual level. The previous RCT was also limited to stroke patients. In addition to stroke, there are many other conditions (such as fractures, lower limb joint replacement, musculoskeletal conditions) require and benefit from rehabilitation. The primary aims of the pilot evaluation study are: (i) To document patient adherence to TR, compared to usual care (ii) To estimate the extent to which TR improves functional status, compared to usual care and (iii) To estimate the cost effectiveness of TR, compared to usual care in eight different health conditions in Singapore.

DETAILED DESCRIPTION:
This is a 12-week quasi-experimental trial of a tele-rehabilitation program involving seven sites and up to 600 adults in Singapore.

ELIGIBILITY:
Inclusion Criteria:

* at least 21 years of age
* Admitted into an inpatient or outpatient rehabilitation unit, nursing home or day care centre for an acute or chronic disability
* Deemed by any members of the multi-disciplinary rehabilitation team to potentially able to safely receive and benefit from rehabilitation post-discharge
* Cognitively able to understand and follow instructions (the Abbreviated Mental Test's score of 6 or above (out of 10).

Exclusion Criteria:

* Patients with previous seizure episodes
* Patients with limb musculoskeletal pain of at least moderate intensity (visual analogue Scale > 6 out of 10)
* Patients with pacemakers.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Adherence to rehabilitation over the course of a 2 week trial period | At 12-weeks post-rehabilitation
  Adherence to the prescribed rehabilitation and exercise therapy will be measured over 12 weeks

SECONDARY OUTCOMES:
EQ-5D | 12-weeks
  Perceived Health Status and Quality of Life
CESD | 12-weeks
  The Center for Epidemiological Studies Depression Scale
IADL | 12-weeks
  The Lawton Instrumental Activities of Daily Living (IADL) Scale
Barthel Index | 12-weeks
  Barthel Index of Activities of Daily Living
Health Service Utilization | 12-weeks
  Use of Health Services over the past three months

CONTACTS AND LOCATIONS:
Overall Officials: Miho Asano, PhD, Principal Investigator — National University of Singapore
Locations (1):
- Miho Asano, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No